CLINICAL TRIAL: NCT04459962
Title: Breath Test Feasibility Trial for Covid-19 Infection Diagnosis
Brief Title: Covid-19 Breath Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ancon Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020ATL01
Record Dates: First submitted 2020-07-03; First posted 2020-07-07 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2020-07

CONDITIONS: Covid-19 Infection
MeSH Terms: conditions — COVID-19 | interventions — Breath Tests

STUDY DESIGN:
Intervention Model Description: Participants who are Covid-19 negative, Covid-19 positive or suspected with Covid-19 infection will be recruited
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): Breath Test and Cheek Swab collection
  Interventions: Diagnostic Test: Breath Test & Cheek Swab

INTERVENTIONS:
Diagnostic Test: Breath Test & Cheek Swab — Breath Sample and Cheek Swab of participants will be used for machine learning (NBT - Nanobiotechnology Biomarkers Tagging) system to develop a profile which can be used later on for Covid-19 Diagnosis.

SUMMARY:
Can Nanotechnology Biomarker Tagging (NBT) be used to detect COVID-19 infection in people presenting for COVID-19 testing?

NBT can be used to detect the substances present in a person's breath. In this study the breath of people presenting for COVID-19 testing is going to be analysed. Analysing a large number of samples from people with COVID-19 (as confirmed by the standard swab test used by the NHS) will enable a breath profile to be produced, ie the substances present in the breath when someone has COVID-19. After the profile has been validated, NBT can be used to test whether or not a person has COVID-19 by seeing if their breath matches the profile.

Using this technology for COVID-19 testing has advantages over the current standard test. The sample can be analysed immediately in the clinical setting and the results are available in 5-10 minutes, so if the person tests negative they can go back to their normal life straight away. The current swab test takes around 72 hours for the results to be available, and the person needs to self-isolate during this time in case they test positive, resulting in potentially unnecessary days of work missed and inconvenience. The breath test is non-invasive and is unlikely to cause any discomfort, as the person is only required to breath normally into the device. This study will also review the practicalities of using this test. It is quick and easy to train people in how to carry out the test, so it could potentially easily be rolled out to testing sites.

DETAILED DESCRIPTION:
This is a Cohort Study which will collect non-invasive, expired breath sample, cheek swab and a Medical and Lifestyle questionnaire from participants.

When the participant presents for COVID-19 testing they will be asked to provide a cheek swab and breath sample, and complete the study questionnaire. They will not need to give any identifiable information or have a second visit. The samples will be analysed immediately and disposed of as clinical waste. ANCON will then use the data to build a breath profile of COVID-19 infection.

Sample and data collection method for inpatients:

* Sequential (daily or every other day as able) breath and swab test will be taken from some of the patients admitted in the hospital (inpatients).
* This will be taken from entry or start of the study to discharge or end of study or until patient or medical staff deem unsuitable to continue
* This will enable to track infection and the relevant profile changes as covid-19 progresses and/or is treated. This will provide vital additional information around identifiers associated with the disease and its progress.

Anonymous Questionnaire - Each participant will be asked questions in the form of a short standard questionnaire based on:

* Medical Information
* Lifestyle Information

ELIGIBILITY:
Inclusion Criteria:

* Male & Females.
* Age Above 16 years old
* All Ethnicity
* Any patients that come for COVID-19 testing
* COVID Negative Patients (Further participants may be selected as control groups who have no current diagnosis of COVID-19.)
* COVID Positive In-Patients

Exclusion Criteria:

* Outside of stated age range - below 16
* Unable to consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
To investigate/ examine the effectiveness of Nanotechnology Biomarker Tagging (NBT) in detecting COVID-19 infection using breath samples of patients with COVID-19 symptoms | 6 Months
  This will be measured by identification of VOCs present in the breath sample of the COVID-19 positive and their relative concentrations compared to a COVID-19 negative breath sample. These will be combined to provide a COVID-19 positive profile

SECONDARY OUTCOMES:
-To profile the unique pattern of Volatile Organic Compounds (VOCs) found in the expired breath of COVID-19 patients using the NBT system (VOC analysis and ML). | 6 months
  This will be measured by identification of VOCs present in the breath sample of the COVID-19 positive and their relative concentrations compared to a COVID-19 negative breath sample using ML. These will be combined to provide a COVID-19 positive profile.
To differentiate this unique profile from the patients that are found to be negative for COVID-19 | 6 months
  The patient samples that return COVID-19 negative will be used as controls for identification of VOCs and relative concentrations that are common to all samples.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Winchester, MBBS, MSc, Principal Investigator — Ashford and St Peter's Hospitals NHS Foundation Trust
Locations (1):
- Ashford and St Peter's Hospitals NHS Foundation Trust, Chertsey, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ajibola OA, Smith D, Spanel P, Ferns GA. Effects of dietary nutrients on volatile breath metabolites. J Nutr Sci. 2013 Oct 31;2:e34. doi: 10.1017/jns.2013.26. eCollection 2013. PMID 25191584
- [Background] Smith D, Spanel P. The challenge of breath analysis for clinical diagnosis and therapeutic monitoring. Analyst. 2007 May;132(5):390-6. doi: 10.1039/b700542n. Epub 2007 Mar 19. PMID 17471381
- [Background] Amann A, Spanel P, Smith D. Breath analysis: the approach towards clinical applications. Mini Rev Med Chem. 2007 Feb;7(2):115-29. doi: 10.2174/138955707779802606. PMID 17305586
- [Background] Gouma PI, Wang L, Simon SR, Stanacevic M. Novel Isoprene Sensor for a Flu Virus Breath Monitor. Sensors (Basel). 2017 Jan 20;17(1):199. doi: 10.3390/s17010199. PMID 28117692
- [Background] Kim, K.-H.Kim., Jahan, S.A., Kabir, E., (2012) A review of breath analysis for diagnosis of human health. TrAC Trends in Analytical Chemistry. v.33, 1-8. https://doi.org/10.1016/j.trac.2011.09.013
- [Background] Lake MA. What we know so far: COVID-19 current clinical knowledge and research. Clin Med (Lond). 2020 Mar;20(2):124-127. doi: 10.7861/clinmed.2019-coron. Epub 2020 Mar 5. PMID 32139372
- [Background] Marczin N, Kharitonov S (2003) Lung Biology in Health and Disease. Disease Markers in Exhaled Breath Edited by: New York: Marcel Dekker; 2003.
- [Background] NHS-England, (2020) Guidance and standard operating procedure COVID-19 virus testing in NHS laboratories.
- [Background] Sethi S, Nanda R, Chakraborty T. Clinical application of volatile organic compound analysis for detecting infectious diseases. Clin Microbiol Rev. 2013 Jul;26(3):462-75. doi: 10.1128/CMR.00020-13. PMID 23824368
- [Background] Risby T., (2005): Current status of clinical breath analysis. In Breath Analysis for Clinical Diagnosis and Therapeutic Monitoring Edited by: Amann A, Smith D. Singapore: World Scientific; 2005:251-265.